CLINICAL TRIAL: NCT05890911
Title: The Importance of Dopamine and Selected Polymorphisms Within the Genes of the Dopaminergic Pathway in Assessment of the Risk of Development and Severity of Sleep Breathing Disorders.
Brief Title: The Meaning of Dopaminergic Pathway in Sleep Breathing Disorders.
Status: Enrolling by invitation | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Joanna Smardz, Principal Investigator, Wroclaw Medical University
Other Study IDs: WMU2/2023
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Sleep Apnea; Sleep-Disordered Breathing
Keywords: sleep apnea; sleep-disordered breathing; sleep disorder; dopamine
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Wake Disorders | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Participants with the diagnosis of sleep-disordered breathing
  Interventions: Diagnostic Test: Polysomnography; Diagnostic Test: Blood dopamine level measurement; Diagnostic Test: Genetical test
- Control group: Healthy participants without diagnosis of sleep-disordered breathing
  Interventions: Diagnostic Test: Polysomnography; Diagnostic Test: Blood dopamine level measurement; Diagnostic Test: Genetical test

INTERVENTIONS:
Diagnostic Test: Polysomnography — Each of the patients will undergo polysomnography
Diagnostic Test: Blood dopamine level measurement — In each of the patients blood dopamine level will be measured
Diagnostic Test: Genetical test — Each of the patients will undergo genetical test focusing on selected single nucleotide polymorphisms within genes regulating the concentration of dopamine - the gene responsible for production of the enzyme catechol-O-methyltransferase (COMT) - rs4680 and rs6269 and genes encoding receptors dopamine (DRD1 - rs686, rs5327 and DRD2 - rs1800497).

SUMMARY:
The participants in the study will be adult patients with suspected sleep-disordered breathing. A one-night polysomnography will be performed using the NOXA1 device (NOX Medical, Reykjavík, Iceland). During the polysomnographic examination, sleep, breathing, heart rate and activity of the masticatory muscles will be recorded. Blood sample will be taken from each of the participants qualified to the study and control group to determine the level of dopamine and used to perform genetic tests of selected single nucleotide polymorphisms occurring within the genes regulating the concentration of dopamine and genes encoding dopamine receptors.

DETAILED DESCRIPTION:
Sleep-disordered breathing (SDB) refers to a spectrum of abnormalities related to sleep. Obstructive sleep apnea (OSA) is the most common type of SDB and affects approximately one billion adults worldwide. Untreated OSA leads to significant comorbidities and increased mortality due to significantly increased risk of stroke and heart attack. Because of limited access to objective sleep studies and the fact that untreated OSA is a real risk factor premature death, the determination of possible organic reasons for its occurrence is a key aspect. The purpose of the study is to determine the importance of dopamine levels and selected single nucleotide polymorphisms within genes regulating the concentration of dopamine - the gene responsible for production of the enzyme catechol-O-methyltransferase (COMT) - rs4680 and rs6269 and genes encoding receptors dopamine (DRD1 - rs686, rs5327 and DRD2 - rs1800497) in assessment of the risk of development and advancement of SDB. The participants of the study will be adult patients hospitalized in the Department of Internal Diseases, Occupational Diseases, Hypertension and Clinical Oncology of the Wroclaw Medical University due to suspicion of SDB. One-night polysomnography study will be performed using the NOXA1 device (NOX Medical, Reykjavík, Iceland) at the Sleep Laboratory. During the examination parameters regarding sleep, breathing, heart rate and activity of the masticatory muscles will be recorded. The study group will consist of the participants in whom, on the basis of 3rd edition of the International Classification of Sleep Disorders of the American Academy of Sleep Medicine SDB will be recognized. Control group will consist of healthy participants matched in terms of age and sex. A blood sample will be collected from all participants to determine the level of dopamine and to perform genetic test of selected single nucleotide polymorphisms within the genes regulating the concentration of dopamine - the gene responsible for production the enzyme catechol-O-methyltransferase (COMT) - rs4680 and rs6269 and genes encoding dopamine receptors (DRD1 - rs686, rs5327 and DRD2 - rs1800497). Study group and control group will be compared and the results will be statistically analysed.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years old
* suspicion of sleep-disordered breathing

Exclusion Criteria:

* age under 18
* age over 80
* severe disorders and systemic diseases (including genetical disorders)
* neurological disorders
* active inflammations
* active cancer
* severe mental disorders and retardation (including genetical)
* taking drugs that could falsify polysomnography
* confirmed alcoholism
* drug addiction
* pregnancy and breast feeding
* treatment using or dependence on any painkillers and/or drugs and substances that may affect nervous, muscular and respiratory system functions
* lack of consent to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion of sleep-disordered breathing referred to the Department of Internal Medicine, Occupational Diseases, Hypertension and Clinical Oncology operating at the Wroclaw Medical University. Healthy controls.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Relationship between sleep-disordered breathing and blood dopamine level. | June 1, 2023 - December 31, 2023
  Each participant will undergo blood test focusing on the level of dopamine.

SECONDARY OUTCOMES:
Relationship between sleep-disordered breathing and polymorphism within genes regulating the concentration and encoding receptors of dopamine. | June 1, 2023 - December 31, 2023
  Each participant will undergo genetical blood test focusing on the polymorphisms within genes regulating the concentration of dopamine - the gene responsible for production of the enzyme catechol-O-methyltransferase (COMT) - rs4680 and rs6269 and genes encoding receptors dopamine (DRD1 - rs686, rs5327 and DRD2 - rs1800497).

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Smardz, Ph.D, Principal Investigator — Wroclaw Medical University
Locations (1):
- Wroclaw Medical Uniwesity, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided